CLINICAL TRIAL: NCT01416571
Title: Immunogenicity and Safety Study of GSK Biologicals' Monovalent Pandemic H5N1 Vaccine 1557484A in Adults Aged 18 - 64 Years
Brief Title: Immunogenicity and Safety Study of GlaxoSmithKline (GSK) Biologicals' Monovalent Pandemic H5N1 Vaccine in Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 112691
Record Dates: First submitted 2011-08-12; First posted 2011-08-15 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2018-09-21 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: H5N1; Influenza vaccine; influenza infection; GSK1557484A
MeSH Terms: conditions — Influenza, Human

ARMS (1):
- Influenza A (H5N1) Group (Experimental): Healthy subjects aged between 18 and 64 years at the time of vaccination received two doses of the Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted, at Day 0 and Day 21. The vaccine was administered intramuscularly in the deltoid region of the arm.
  Interventions: Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus Monovalent Vaccine, Adjuvanted — Intramuscular (IM), two doses

SUMMARY:
This trial will assess the immunogenicity and safety of GSK Biologicals' vaccine GSK1557484A, prepared from old concentrated monobulk material, in adults aged 18 to 64 years, when administered up to 5 years following production.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol.
* A male or female 18 to 64 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Stable general health as established by medical history and clinical examination before entering into the study.
* Subject access to a consistent means of telephone contact, land line or mobile, but NOT a pay phone or other multiple-user device.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Previous vaccination at any time with an H5N1 vaccine.
* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Presence of significant acute or chronic, uncontrolled medical or psychiatric illness.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the potential subject unable/unlikely to provide accurate safety reports.
* Presence of a temperature ≥ 38.0ºC, or acute symptoms greater than "mild" severity on the scheduled date of first dose.
* Diagnosed with cancer, or treatment for cancer, within 3 years.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Receipt of systemic glucocorticoids within 1 month prior to study enrolment, or any other cytotoxic or immunosuppressive drug within 6 months of study enrolment. Topical, intra-articularly injected, or inhaled glucocorticoids, topical calcineurin inhibitors or imiquimod are allowed.
* Receipt of any immunoglobulins and/or any blood products within 3 months before first study vaccination or planned administration of any of these products during the study period.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin. Persons receiving individual doses of low molecular weight heparin outside of 24 hours prior to dosing, are eligible. Persons receiving prophylactic antiplatelet medications, and without a clinically-apparent bleeding tendency, are eligible.
* An acute evolving neurological disorder or history of Guillain-Barré syndrome within 6 weeks of receipt of seasonal influenza vaccine.
* Administration of an inactivated or a live, attenuated seasonal influenza vaccine within 14 days before the first study vaccine dose, or of any other vaccine(s) not foreseen by the study protocol within 30 days before the first study vaccine dose.
* Planned administration of any vaccine(s) not foreseen by the study protocol through completion of the Day 42 visit.
* Any known or suspected allergy to any constituent of influenza vaccines, or history of severe reaction to a previous influenza vaccination.
* Known pregnancy or a positive urine beta-human chorionic gonadotropin test result prior to the first study vaccine dose.
* Lactating or nursing women.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2011-08-12; Primary Completion 2011-11-29 (Actual); Study Completion 2012-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Godeaux O, Izurieta P, Madariaga M, Drame M, Li P, Vaughn DW. Immunogenicity and safety of AS03A-adjuvanted H5N1 influenza vaccine prepared from bulk antigen after stockpiling for 4 years. Vaccine. 2015 Apr 27;33(18):2189-95. doi: 10.1016/j.vaccine.2014.07.062. Epub 2014 Jul 30. PMID 25090645
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 112691 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in two phases: the Primary Vaccination Phase (up to Day 84) and the Immunogenicity and Safety follow-up Phase (up to Day 385).
Period: Overall Study
Arm/Group | Influenza A (H5N1) Group
Started | 78
Completed | 76 (Number of subjects completed at Day 385.)
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (13.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects Against the H5N1 Strain of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination reciprocal HI titer less than (<) 1:10 and a post-vaccination reciprocal HI titer greater than or equal to (≥) 1:40 or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a four-fold increase in post-vaccination reciprocal titer against the vaccine virus.
Time Frame: At Day 42
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity at Day 42, which included all evaluable subjects who received the study vaccine doses and for whom the assay results for antibodies against vaccine-homologous H5N1 Hemagglutinin (HA) antigen for the blood samples taken at Day 0, and Day 42 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 75
Participants | 72

2. Primary Outcome: Mean Geometric Increase (MGI) for the H5N1 Strain of Influenza Disease.
Description: MGI was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer for the vaccine virus.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 75
ratio | 41.7 [32.0 to 54.3]

3. Primary Outcome: Number of Seroprotected Subjects Against the H5N1 Strain of Influenza Disease.
Description: A seroprotected subject was defined as a vaccinated subject who had H5N1 reciprocal HI titers ≥ 1:40 against the vaccine-homologous virus.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 75
Participants | 74

4. Secondary Outcome: Number of Seropositive Subjects Against the H5N1 Strain of Influenza Disease.
Description: A seropositive subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:10.
Time Frame: At Day 0 and Day 42
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 75
Participants
  H5N1 at Day 0 | 26
  H5N1 at Day 42 | 75

5. Secondary Outcome: Titers for Serum HI Antibodies Against the H5N1 Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 0 and Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 75
titers
  H5N1 at Day 0 | 7.5 [6.5 to 8.6]
  H5N1 at Day 42 | 311.3 [249.2 to 389.0]

6. Secondary Outcome: Number of Seropositive Subjects Against the H5N1 Strain of Influenza Disease.
Description: A seropositive subject was defined as a vaccinated subject who had a serum HI titer ≥ 1:10.
Time Frame: At Day 0 and Day 182
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for persistence at Day 182, which included all evaluable subjects who received the study vaccine doses and for whom the assay results for antibodies against the vaccine-homologous H5N1 HA antigen for the blood samples taken at Day 0 and Day 182 were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 74
Participants
  H5N1 at Day 0 | 27
  H5N1 at Day 182: number analyzed (Participants) | 73
  H5N1 at Day 182 | 73

7. Secondary Outcome: Titers for Serum HI Antibodies Against the H5N1 Strain of Influenza Disease.
Description: Titers are presented as geometric mean titers (GMTs).
Time Frame: At Day 0 and Day 182
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 74
titers
  H5N1 at Day 0 | 7.8 [6.6 to 9.1]
  H5N1 at Day 182: number analyzed (Participants) | 73
  H5N1 at Day 182 | 56.3 [47.0 to 67.5]

8. Secondary Outcome: Number of Seroprotected Subjects Against the H5N1 Strain of Influenza Disease.
Description: as for outcome 3
Time Frame: At Day 0 and Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 74
Participants
  H5N1 at Day 0 | 3
  H5N1 at Day 182: number analyzed (Participants) | 73
  H5N1 at Day 182 | 56

9. Secondary Outcome: Number of Seroconverted Subjects Against the H5N1 Strain of Influenza Disease.
Description: A seroconverted subject was defined as a vaccinated subject who had either a pre-vaccination reciprocal HI titer < 1:10 and a post-vaccination reciprocal HI titer (≥) 1:40 or a pre-vaccination reciprocal HI titer ≥ 1:10 and at least a four-fold increase in post-vaccination reciprocal titer against the vaccine virus.
Time Frame: At Day 182
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 73
Participants | 48

10. Secondary Outcome: Mean Geometric Increase (MGI) for the H5N1 Strain of Influenza Disease.
Description: as for outcome 2
Time Frame: At Day 182
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 73
ratio | 7.2 [5.8 to 9.0]

11. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of any solicited local symptoms regardless of intensity grade. Grade 3 pain = significant pain at rest; prevented normal activities. Grade 3 Redness/Swelling = Redness/Swelling >100 millimeters (mm).
Time Frame: During the 7-day follow-up period (Days 0-6) after any vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any Pain | 71
  Any Redness | 7
  Any Swelling | 12
  Grade 3 Pain | 6
  Grade 3 Redness | 0
  Grade 3 Swelling | 0

12. Secondary Outcome: Duration of Solicited Local Symptoms After Vaccination.
Description: Assessed solicited local symptoms were pain, redness and swelling. Duration was defined as the number of days with any grade of local symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects who received at least one study vaccination, on subjects who experienced the specific symptom.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 70
days
  Pain, Dose 1 | 3.0 [2.0 to 4.0]
  Pain, Dose 2: number analyzed (Participants) | 60
  Pain, Dose 2 | 3.0 [2.0 to 3.0]
  Redness, Dose1: number analyzed (Participants) | 5
  Redness, Dose1 | 2.0 [1.0 to 2.0]
  Redness, Dose 2: number analyzed (Participants) | 3
  Redness, Dose 2 | 3.0 [1.0 to 4.0]
  Swelling, Dose 1: number analyzed (Participants) | 10
  Swelling, Dose 1 | 2.0 [1.0 to 3.0]
  Swelling, Dose 2: number analyzed (Participants) | 5
  Swelling, Dose 2 | 1.0 [1.0 to 2.0]

13. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache, joint pain at other location (joint pain), muscle aches, shivering, sweating and fever. Any = occurrence of any solicited general symptoms regardless of intensity grade or relationship to vaccination. Any fever was defined as axillary temperature ≥ 38 degrees Celsius (°C). Grade 3 = general symptom that prevented normal activities. Grade 3 fever = fever ≥ 39.0°C. Related = general symptom assessed by the investigator as causally related to the vaccination.
Time Frame: During the 7-day follow-up period (Days 0-6) after any vaccination
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any Fatigue | 35
  Grade 3 Fatigue | 3
  Related Fatigue | 26
  Any Gastrointestinal | 13
  Grade 3 Gastrointestinal | 0
  Related Gastrointestinal | 6
  Any Headache | 28
  Grade 3 Headache | 1
  Related Headache | 20
  Any Joint Pain | 13
  Grade 3 Joint Pain | 0
  Related Joint Pain | 13
  Any Muscle Aches | 31
  Grade 3 Muscle Aches | 3
  Related Muscle Aches | 27
  Any Shivering | 10
  Grade 3 Shivering | 1
  Related Shivering | 10
  Any Sweating | 11
  Grade 3 Sweating | 0
  Related Sweating | 8
  Any Fever | 0
  Grade 3 Fever | 0
  Related Fever | 0

14. Secondary Outcome: Duration of Solicited General Symptoms After Vaccination.
Description: Assessed solicited general symptoms were fatigue, gastrointestinal, headache, joint pain at other location (joint pain), muscle aches, increased sweating and shivering. Duration was defined as the number of days with any grade of general symptoms.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose
Population: as for outcome 12
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 26
days
  Fatigue, Dose 1: number analyzed (Participants) | 23
  Fatigue, Dose 1 | 2.0 [1.0 to 3.0]
  Fatigue, Dose 2 | 2.0 [1.0 to 3.0]
  Gastrointestinal, Dose 1: number analyzed (Participants) | 11
  Gastrointestinal, Dose 1 | 2.0 [1.0 to 3.0]
  Gastrointestinal, Dose 2: number analyzed (Participants) | 7
  Gastrointestinal, Dose 2 | 2.0 [2.0 to 3.0]
  Headache, Dose 1: number analyzed (Participants) | 20
  Headache, Dose 1 | 1.5 [1.0 to 2.0]
  Headache, Dose 2: number analyzed (Participants) | 18
  Headache, Dose 2 | 1.5 [1.0 to 2.0]
  Joint Pain, Dose 1: number analyzed (Participants) | 6
  Joint Pain, Dose 1 | 1.5 [1.0 to 3.0]
  Joint Pain, Dose 2: number analyzed (Participants) | 12
  Joint Pain, Dose 2 | 2.0 [1.5 to 3.0]
  Muscle aches, Dose 1: number analyzed (Participants) | 18
  Muscle aches, Dose 1 | 2.0 [1.0 to 3.0]
  Muscle aches, Dose 2: number analyzed (Participants) | 24
  Muscle aches, Dose 2 | 2.0 [1.0 to 2.5]
  Increased sweating, Dose 1: number analyzed (Participants) | 7
  Increased sweating, Dose 1 | 2.0 [1.0 to 3.0]
  Increased sweating, Dose 2: number analyzed (Participants) | 6
  Increased sweating, Dose 2 | 2.5 [1.0 to 3.0]
  Shivering, Dose 1: number analyzed (Participants) | 2
  Shivering, Dose 1 | 2.0 [1.0 to 3.0]
  Shivering, Dose 2: number analyzed (Participants) | 9
  Shivering, Dose 2 | 1.0 [1.0 to 1.0]

15. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Attended Adverse Events (MAEs).
Description: MAE was defined as any unsolicited symptom that received medical attention such as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any = occurrence of any MAEs regardless of intensity grade or relationship to vaccination. Grade 3 = event which prevented normal activities Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 to Day 84
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any MAEs | 20
  Grade 3 MAEs | 6
  Related MAEs | 0

16. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Medically Attended Adverse Events (MAEs).
Description: MAE was defined as any unsolicited symptom that received medical attention such as hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel for any reason. Any = occurrence of any MAEs regardless of intensity grade or relationship to vaccination. Grade 3 = event which prevented normal activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 to Day 385
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any MAEs | 49
  Grade 3 MAEs | 9
  Related MAEs | 0

17. Secondary Outcome: Number of Subjects With Potential Immune Mediated Disease (s) (pIMDs).
Description: pIMDs are a subset of AEs that include both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 to Day 84 and from Day 0 to Day 385
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  pIMD(s), Day 0 to Day 84 | 0
  pIMD(s), Day 0 to Day 385 | 0

18. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical and Haematological Parameters.
Description: Assessed biochemical and haematological parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), blood urea nitrogen (BUN), creatinine (CREA), eosinophils (EOS), haematocrit (HCRIT), haemoglobin (HBIN), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC), total bilirubin (Total BIR), bilirubin conjugated/direct (BIL con/dir). Per parameter, it was assessed whether subjects had laboratory values unknown, below, within or above the normal ranges. This outcome presents BAS, EOS and HCRIT results.
Time Frame: At Day 0 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  BAS, unknown, Day 0 | 1
  BAS, unknown, Day 42: number analyzed (Participants) | 77
  BAS, unknown, Day 42 | 1
  BAS, below, Day 0 | 0
  BAS, below, Day 42: number analyzed (Participants) | 77
  BAS, below, Day 42 | 0
  BAS, within, Day 0 | 77
  BAS, within, Day 42: number analyzed (Participants) | 77
  BAS, within, Day 42 | 76
  BAS, above, Day 0 | 0
  BAS, above, Day 42: number analyzed (Participants) | 77
  BAS, above, Day 42 | 0
  EOS, unknown, Day 0 | 1
  EOS, unknown, Day 42: number analyzed (Participants) | 77
  EOS, unknown, Day 42 | 1
  EOS, below, Day 0 | 23
  EOS, below, Day 42: number analyzed (Participants) | 77
  EOS, below, Day 42 | 12
  EOS, within, Day 0 | 53
  EOS, within, Day 42: number analyzed (Participants) | 77
  EOS, within, Day 42 | 64
  EOS, above, Day 0 | 1
  EOS, above, Day 42: number analyzed (Participants) | 77
  EOS, above, Day 42 | 0
  HCRIT, unknown, Day 0 | 0
  HCRIT, unknown, Day 42: number analyzed (Participants) | 77
  HCRIT, unknown, Day 42 | 1
  HCRIT, below, Day 0 | 2
  HCRIT, below, Day 42: number analyzed (Participants) | 77
  HCRIT, below, Day 42 | 5
  HCRIT, within, Day 0 | 68
  HCRIT, within, Day 42: number analyzed (Participants) | 77
  HCRIT, within, Day 42 | 66
  HCRIT, above, Day 0 | 8
  HCRIT, above, Day 42: number analyzed (Participants) | 77
  HCRIT, above, Day 42 | 5

19. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical and Haematological Parameters.
Description: Assessed biochemical and haematological parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), blood urea nitrogen (BUN), creatinine (CREA), eosinophils (EOS), haematocrit (HCRIT), haemoglobin (HBIN), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC), total bilirubin (Total BIR), bilirubin conjugated/direct (BIL con/dir). Per parameter, it was assessed whether subjects had laboratory values unknown, below, within or above the normal ranges. This outcome presents HBIN, LYM and MON results.
Time Frame: At Day 0 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  HBIN, unknown, Day 0 | 0
  HBIN, unknown, Day 42: number analyzed (Participants) | 77
  HBIN, unknown, Day 42 | 1
  HBIN, below, Day 0 | 7
  HBIN, below, Day 42: number analyzed (Participants) | 77
  HBIN, below, Day 42 | 6
  HBIN, within, Day 0 | 68
  HBIN, within, Day 42: number analyzed (Participants) | 77
  HBIN, within, Day 42 | 68
  HBIN, above, Day 0 | 3
  HBIN, above, Day 42: number analyzed (Participants) | 77
  HBIN, above, Day 42 | 2
  LYM, unknown, Day 0 | 1
  LYM, unknown, Day 42: number analyzed (Participants) | 77
  LYM, unknown, Day 42 | 1
  LYM, below, Day 0 | 2
  LYM, below, Day 42: number analyzed (Participants) | 77
  LYM, below, Day 42 | 0
  LYM, within, Day 0 | 75
  LYM, within, Day 42: number analyzed (Participants) | 77
  LYM, within, Day 42 | 76
  LYM, above, Day 0 | 0
  LYM, above, Day 42: number analyzed (Participants) | 77
  LYM, above, Day 42 | 0
  MON, unknown, Day 0 | 1
  MON, unknown, Day 42: number analyzed (Participants) | 77
  MON, unknown, Day 42 | 1
  MON, below, Day 0 | 46
  MON, below, Day 42: number analyzed (Participants) | 77
  MON, below, Day 42 | 9
  MON, within, Day 0 | 31
  MON, within, Day 42: number analyzed (Participants) | 77
  MON, within, Day 42 | 67
  MON, above, Day 0 | 0
  MON, above, Day 42: number analyzed (Participants) | 77
  MON, above, Day 42 | 0

20. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical and Haematological Parameters.
Description: Assessed biochemical and haematological parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), blood urea nitrogen (BUN), creatinine (CREA), eosinophils (EOS), haematocrit (HCRIT), haemoglobin (HBIN), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC), total bilirubin (Total BIR), bilirubin conjugated/direct (BIL con/dir). Per parameter, it was assessed whether subjects had laboratory values unknown, below, within or above the normal ranges. This outcome presents NEU, PLA and RBC results.
Time Frame: At Day 0 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  NEU, unknown, Day 0 | 1
  NEU, unknown, Day 42: number analyzed (Participants) | 77
  NEU, unknown, Day 42 | 1
  NEU, below, Day 0 | 2
  NEU, below, Day 42: number analyzed (Participants) | 77
  NEU, below, Day 42 | 1
  NEU, within, Day 0 | 71
  NEU, within, Day 42: number analyzed (Participants) | 77
  NEU, within, Day 42 | 75
  NEU, above, Day 0 | 4
  NEU, above, Day 42: number analyzed (Participants) | 77
  NEU, above, Day 42 | 0
  PLA, unknown, Day 0 | 3
  PLA, unknown, Day 42: number analyzed (Participants) | 77
  PLA, unknown, Day 42 | 2
  PLA, below, Day 0 | 0
  PLA, below, Day 42: number analyzed (Participants) | 77
  PLA, below, Day 42 | 1
  PLA, within, Day 0 | 74
  PLA, within, Day 42: number analyzed (Participants) | 77
  PLA, within, Day 42 | 74
  PLA, above, Day 0 | 1
  PLA, above, Day 42: number analyzed (Participants) | 77
  PLA, above, Day 42 | 0
  RBC, unknown, Day 0 | 0
  RBC, unknown, Day 42: number analyzed (Participants) | 77
  RBC, unknown, Day 42 | 1
  RBC, below, Day 0 | 5
  RBC, below, Day 42: number analyzed (Participants) | 77
  RBC, below, Day 42 | 3
  RBC, within, Day 0 | 72
  RBC, within, Day 42: number analyzed (Participants) | 77
  RBC, within, Day 42 | 72
  RBC, above, Day 0 | 1
  RBC, above, Day 42: number analyzed (Participants) | 77
  RBC, above, Day 42 | 1

21. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical and Haematological Parameters.
Description: Assessed biochemical and haematological parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), blood urea nitrogen (BUN), creatinine (CREA), eosinophils (EOS), haematocrit (HCRIT), haemoglobin (HBIN), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC), total bilirubin (Total BIR), bilirubin conjugated/direct (BIL con/dir). Per parameter, it was assessed whether subjects had laboratory values unknown, below, within or above the normal ranges. This outcome presents WBC, ALT and AST results.
Time Frame: At Day 0 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  WBC, unknown, Day 0 | 1
  WBC, unknown, Day 42: number analyzed (Participants) | 77
  WBC, unknown, Day 42 | 1
  WBC, below, Day 0 | 2
  WBC, below, Day 42: number analyzed (Participants) | 77
  WBC, below, Day 42 | 2
  WBC, within, Day 0 | 72
  WBC, within, Day 42: number analyzed (Participants) | 77
  WBC, within, Day 42 | 74
  WBC, above, Day 0 | 3
  WBC, above, Day 42: number analyzed (Participants) | 77
  WBC, above, Day 42 | 0
  ALT, unknown, Day 0 | 0
  ALT, unknown, Day 42: number analyzed (Participants) | 77
  ALT, unknown, Day 42 | 2
  ALT, below, Day 0 | 0
  ALT, below, Day 42: number analyzed (Participants) | 77
  ALT, below, Day 42 | 0
  ALT, within, Day 0 | 76
  ALT, within, Day 42: number analyzed (Participants) | 77
  ALT, within, Day 42 | 73
  ALT, above, Day 0 | 2
  ALT, above, Day 42: number analyzed (Participants) | 77
  ALT, above, Day 42 | 2
  AST, unknown, Day 0 | 0
  AST, unknown, Day 42: number analyzed (Participants) | 77
  AST, unknown, Day 42 | 2
  AST, below, Day 0 | 0
  AST, below, Day 42: number analyzed (Participants) | 77
  AST, below, Day 42 | 0
  AST, within, Day 0 | 78
  AST, within, Day 42: number analyzed (Participants) | 77
  AST, within, Day 42 | 74
  AST, above, Day 0 | 0
  AST, above, Day 42: number analyzed (Participants) | 77
  AST, above, Day 42 | 1

22. Secondary Outcome: Number of Subjects With Normal and Abnormal Biochemical and Haematological Parameters.
Description: Assessed biochemical and haematological parameters were alanine aminotransferase (ALT), aspartate aminotransferase (AST), basophils (BAS), blood urea nitrogen (BUN), creatinine (CREA), eosinophils (EOS), haematocrit (HCRIT), haemoglobin (HBIN), lymphocytes (LYM), monocytes (MON), neutrophils (NEU), platelets (PLA), red blood cells (RBC), white blood cells (WBC), total bilirubin (Total BIL), bilirubin conjugated/direct (BIL con/dir). Per parameter, it was assessed whether subjects had laboratory values unknown, below, within or above the normal ranges. This outcome presents Total BIL, BIL con/dir, CREA and BUN results.
Time Frame: At Day 0 and Day 42
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Total BIL, unknown, Day 0 | 0
  Total BIL, unknown, Day 42: number analyzed (Participants) | 77
  Total BIL, unknown, Day 42 | 2
  Total BIL, below, Day 0 | 0
  Total BIL, below, Day 42: number analyzed (Participants) | 77
  Total BIL, below, Day 42 | 0
  Total BIL, within, Day 0 | 76
  Total BIL, within, Day 42: number analyzed (Participants) | 77
  Total BIL, within, Day 42 | 74
  Total BIL, above, Day 0 | 2
  Total BIL, above, Day 42: number analyzed (Participants) | 77
  Total BIL, above, Day 42 | 1
  BIL con/dir, unknown, Day 0 | 0
  BIL con/dir, unknown, Day 42: number analyzed (Participants) | 77
  BIL con/dir, unknown, Day 42 | 2
  BIL con/dir, below, Day 0 | 0
  BIL con/dir, below, Day 42: number analyzed (Participants) | 77
  BIL con/dir, below, Day 42 | 0
  BIL con/dir, within, Day 0 | 78
  BIL con/dir, within, Day 42: number analyzed (Participants) | 77
  BIL con/dir, within, Day 42 | 75
  BIL con/dir, above, Day 0 | 0
  BIL con/dir, above, Day 42: number analyzed (Participants) | 77
  BIL con/dir, above, Day 42 | 0
  CREA, unknown, Day 0 | 0
  CREA, unknown, Day 42: number analyzed (Participants) | 77
  CREA, unknown, Day 42 | 2
  CREA, below, Day 0 | 5
  CREA, below, Day 42: number analyzed (Participants) | 77
  CREA, below, Day 42 | 5
  CREA, within, Day 0 | 73
  CREA, within, Day 42: number analyzed (Participants) | 77
  CREA, within, Day 42 | 68
  CREA, above, Day 0 | 0
  CREA, above, Day 42: number analyzed (Participants) | 77
  CREA, above, Day 42 | 2
  BUN, unknown, Day 0 | 0
  BUN, unknown, Day 42: number analyzed (Participants) | 77
  BUN, unknown, Day 42 | 2
  BUN, below, Day 0 | 1
  BUN, below, Day 42: number analyzed (Participants) | 77
  BUN, below, Day 42 | 0
  BUN, within, Day 0 | 76
  BUN, within, Day 42: number analyzed (Participants) | 77
  BUN, within, Day 42 | 74
  BUN, above, Day 0 | 1
  BUN, above, Day 42: number analyzed (Participants) | 77
  BUN, above, Day 42 | 1

23. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = occurrence of an unsolicited AE regardless of intensity grade or relationship to vaccination. Grade 3 = event which prevented normal activities. Related = event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 to Day 20 and from Day 0 to Day 84.
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any unsolicited AEs [Days 0-20] | 38
  Grade 3 unsolicited AEs [Days 0-20] | 5
  Related unsolicited AEs [Days 0-20] | 7
  Any unsolicited AEs [Days 0-84] | 46
  Grade 3 unsolicited AEs [Days 0-84] | 7
  Related unsolicited AEs [Days 0-84] | 7

24. Secondary Outcome: Number of Subjects With Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) was defined as any untoward medical occurrence that resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or resulted in a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: From Day 0 to Day 84 and from Day 0 to Day 385
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Influenza A (H5N1) Group
Number analyzed (Participants) | 78
Participants
  Any SAEs [Days 0-84] | 2
  Any SAEs [Days 0-385] | 3
  Related SAEs [Days 0-84] | 0
  Related SAEs [Days 0-385] | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: Within the 7-day period after primary vaccination. Unsolicited AEs: From Day 0 to Day 84. SAEs: from Day 0 to Day 385.
Arm/Group | Influenza A (H5N1) Group
Serious Adverse Events (participants affected / at risk) | 3/78
Other Adverse Events (participants affected / at risk) | 74/78
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) Group (N=78)
Hernia obstructive (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Influenza A (H5N1) Group (N=78)
Pain (General disorders) | 71
Redness (General disorders) | 7
Swelling (General disorders) | 12
Fatigue (General disorders) | 35
Gastrointestinal (General disorders) | 13
Headache (General disorders) | 28
Joint pain (General disorders) | 13
Muscle aches (General disorders) | 31
Shivering (General disorders) | 10
Sweating (General disorders) | 11
Nasopharyngitis (Infections and infestations) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.